CLINICAL TRIAL: NCT04957888
Title: Investigation on the Microbial Biomarkers of AGI in the Early Stage
Brief Title: Microbial Markers for AGI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: LM2020203
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Acute Gastrointestinal Injury
Keywords: microbiome; metabolome; biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training group: the observational group to find out the potential biomarker
  Interventions: Other: none intervention
- validation group: the validation group to validate the parameters used for early diagnosis
  Interventions: Other: none intervention

INTERVENTIONS:
Other: none intervention — none intervention.

SUMMARY:
AGI is very common in ICU and sometimes will trigger the development of gut derived sepsis. Thus, to find out the biomarker in early stage is very important to improve the overall prognosis of critically ill patients. In this project we try to find out the microbial biomarker of AGI through multi-omic technology.

ELIGIBILITY:
Inclusion Criteria: All those critically ill patients with anticipated ICU stay for more than 2 days Exclusion Criteria:Patients will be excluded if they have any of the following situations: patients who have not signed the informed consent; Unable to tolerate intra-abdominal pressure monitoring; pregnant woman; Patients after bladder surgery; Systemic diseases and recent use of related drugs; He had a history of infectious diseases, such as tuberculosis or PPD positive. History of hypertension and poor blood pressure control (SBP / DBP > = 140mmHg); Patients with severe mental illness; Long term use of traditional Chinese medicine, probiotics, gastric mucosal protective agents, proton pump inhibitors, chemotherapy or immunosuppressive drugs, etc. were not included if the drug was not stopped within one month before admission.

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: ICU patients
Sampling Method: Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
The AUC value of the combined markers | 1 year
  The combined diagnostic accuracy of AGI through omic parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No